CLINICAL TRIAL: NCT02596893
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Multicenter Study to Investigate the Efficacy and Safety of Mongersen (GED-0301) for the Treatment of Subjects With Active Crohn's Disease
Brief Title: Efficacy and Safety Study of Mongersen (GED-0301) for the Treatment of Subjects With Active Crohn's Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GED-0301-CD-002
Record Dates: First submitted 2015-11-03; First posted 2015-11-04 (Estimated); Results first posted 2019-01-23 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Crohn Disease
Keywords: Crohn's Disease; GED-0301; Mongersen; IBD; Safety; Efficacy
MeSH Terms: conditions — Crohn Disease | interventions — GED0301

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- GED0301 160mg x 12 weeks followed by periodic 160 mg GED0301 (Experimental): GED-0301 160 mg once daily (QD) for 12 weeks; followed by placebo QD for 4 weeks; followed by alternating GED-0301 160 mg QD for 4 weeks and placebo QD for 4 weeks, until the the Week 52 Visit
  Interventions: Drug: GED-0301; Drug: Placebo
- GED0301 160mg x 12 weeks followed by periodic GED0301 40mg (Experimental): GED-0301 160 mg once daily (QD) for 12 weeks; followed by placebo QD for 4 weeks; followed by alternating GED-0301 40 mg QD for 4 weeks and placebo QD for 4 weeks, until the Week 52 Visit
  Interventions: Drug: GED-0301; Drug: Placebo
- GED0301 160mg x 12 weeks followed by continuous GED0301 40mg (Experimental): GED-0301 160 mg once daily (QD) for 12 weeks; followed by continuous GED-0301 40 mg QD, until the Week 52 Visit
  Interventions: Drug: GED-0301
- Placebo (Placebo Comparator): Placebo once daily (QD) until the Week 52 Visit
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GED-0301
  Arms: GED0301 160mg x 12 weeks followed by continuous GED0301 40mg; GED0301 160mg x 12 weeks followed by periodic 160 mg GED0301; GED0301 160mg x 12 weeks followed by periodic GED0301 40mg
Drug: Placebo
  Arms: GED0301 160mg x 12 weeks followed by periodic 160 mg GED0301; GED0301 160mg x 12 weeks followed by periodic GED0301 40mg; Placebo

SUMMARY:
The purpose of study is to test the effects of an experimental medication GED-0301 (mongersen) in patients who have active Crohn's disease. The study will test GED-0301 compared to placebo for 52 weeks. The study treatment is blinded which means that patients and the study doctor will not know which treatment has been assigned. Patients in this study will be allowed treatment with stable doses of oral aminosalicylates, oral corticosteroids, immunosupressants and antibiotics for the treatment of Crohn's disease.

After 12 weeks in the study until the end of the study, patients who do not have an improvement in their Crohns disease symptoms will have the option to enter a long term active treatment study. Participants who discontinued the study anytime or completed the study at Week 52 were then observed for an additional 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

* Male or female ≥ 18 years
* Active Crohn's disease (CD) disease as determined by the Crohn's Disease Activity Index (CDAI) score and the Simple Endoscopic Score for Crohn's Disease (SES-CD)
* Must meet a determined average minimum number of daily stools or rating of abdominal pain over a 7 day period
* Subject must have failed or experienced intolerance to at least one of the following: budesonide; systemic corticosteroids; immunosuppressants (eg, azathiopurine, 6-mercaptopurine, or methotrexate); or biologics for the treatment of CD.

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

* Diagnosis of ulcerative colitis (UC), indeterminate colitis, ischemic colitis, microscopic colitis, radiation colitis or diverticular disease-associated colitis
* Local manifestations of Crohn's Disease (CD) such as symptomatic/severe strictures, abscesses, short bowel syndrome; or other disease complications for which surgery might be indicated or could confound the evaluation of efficacy
* Intestinal resection within 6 months or any intra-abdominal surgery within 3 months prior to the Screening Visit
* Ileostomy or a colostomy
* Subject has a history of any clinically significant medical condition that, in the investigator's opinion, would prevent the subject from participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 701 (Actual)
Dates: Start 2015-12-08 (Actual); Primary Completion 2018-01-05 (Actual); Study Completion 2018-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Rossiter, MD, Study Director — Celgene Corporation
Locations (537):
- United States (150):
  - ADDC Research LLC, Huntsville, Alabama
  - Arizona Digestive Health, Mesa, Arizona
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Colon & Digestive Health Specialists, Scottsdale, Arizona
  - Arizona Digestive Health, Sun City, Arizona
  - Gastroenterology Associates PA, Little Rock, Arkansas
  - HCP Clinical Research LLC, Anaheim, California
  - T. Joseph Raoof MD Inc, Encino, California
  - Valley View Internal Medicine, Garden Grove, California
  - OM Research, Lancaster, California
  - University of Southern California Medical Center, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Facey Medical Foundation, Mission Hills, California
  - Medical Associates Research Group Inc., San Diego, California
  - Clinical Applications Laboratories Inc, San Diego, California
  - University of California at San Francisco, San Francisco, California
  - Ventura Clinical Trials, Ventura, California
  - University Of Colorado, Aurora, Colorado
  - Innovative Clinical Research, Lafayette, Colorado
  - Connecticut Gastroenterology Institute, Bristol, Connecticut
  - Medical Research Center of Connecticut LLC, Hamden, Connecticut
  - Connecticut GI PC Research Division, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Florida Medical Research - Southeastern Integrated Medical, Gainesville, Florida
  - Sarkis Clinical Trials - Parent, Gainesville, Florida
  - Borland-Groover Clinic, Jacksonville, Florida
  - Florida Center for Gastroenterology, Largo, Florida
  - Advance Medical Research Center, Miami, Florida
  - Cordova Research Institute, Miami, Florida
  - My Community Research Center inc, Miami, Florida
  - Sanitas Research, Miami, Florida
  - Galiz Research LLC, Miami Springs, Florida
  - Gastroenterology Group of Naples, Naples, Florida
  - GCRM, Orlando, Florida
  - Center For Digestive Health, Orlando, Florida
  - BRCR Medical Center Inc., Plantation, Florida
  - Advanced Medical Research Center, Port Orange, Florida
  - East Coast Institute for Research LLC, Saint Augustine, Florida
  - Cleveland Clinic Florida Weston, Weston, Florida
  - Shafran Gastroenterology Center, Winter Park, Florida
  - Atlanta Gastroenterology Associates, LLC, Atlanta, Georgia
  - Georgia Regents University, Augusta, Georgia
  - Columbus Regional Research Institute, Columbus, Georgia
  - Atlanta Gastroenterology Specialists PC, Suwanee, Georgia
  - Grand Teton Research Group PLLC, Idaho Falls, Idaho
  - Northwestern University-Feinberg School of Medicine, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - NorthShore University HealthSystem, Highland Park, Illinois
  - Indiana University, Indianapolis, Indiana
  - Iowa Digestive Disease Center, Clive, Iowa
  - Health Science Research Center, LLC, Pratt, Kansas
  - Heartland Research Associates LLC, Wichita, Kansas
  - Via Christi Research a division of Via Christi Hospitals Wichita Inc, Wichita, Kansas
  - Graves Gilbert Clinic, Bowling Green, Kentucky
  - University of Kentucky Medical Center, Lexington, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Gastroenterology Associates LLC, Baton Rouge, Louisiana
  - Clinical Trials of SW Louisiana LLC, Lake Charles, Louisiana
  - Louisiana Research Center LLC, Shreveport, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Metropolitan Gastroenterology, Chevy Chase, Maryland
  - Gastro Center of Maryland, Columbia, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Commonwealth Clinical Studies PLLC, Brockton, Massachusetts
  - UMass Medical Center, Worcester, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Medex Research Institute, Caro, Michigan
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Henry Ford Medical Center - New Center One, Novi, Michigan
  - Gastroenterology Associates of Western Michigan PLC, Wyoming, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Ehrhardt Clinical Research LLC, Belton, Missouri
  - Jefferson City Medical Group, Jefferson City, Missouri
  - Mercy Research, Springfield, Missouri
  - Saint Louis University, St Louis, Missouri
  - Mercy Clinic East Communities d/b/a Mercy Health Research, Washington, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - AGA Clinical Research Associates LLC, Egg Harbor, New Jersey
  - Southwest Gastroenterology Associates PC, Albuquerque, New Mexico
  - Sing Chan Private Practice, Flushing, New York
  - NYU Langone Nassau Gastroenterology Associates, Great Neck, New York
  - Montefiore Medical Center PRIME, Lake Success, New York
  - The Feinstein Institute for Medical Research PRIME, Manhasset, New York
  - Winthrop University Hospital, Mineola, New York
  - North Shore Long Island Jewish Health System, New Hyde Park, New York
  - Concord Medical Group PRIME, New York, New York
  - New York University School of Medicine, New York, New York
  - New York - Presbyterian/Weill Cornell Medical Center, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - Premier Medical Group of the Hudson Valley PC, Poughkeepsie, New York
  - University of Rochester, Rochester, New York
  - Asheville Gastroenterology Associates, PA, Asheville, North Carolina
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Carolina Center for Liver Disease, Charlotte, North Carolina
  - Gaffney Health Services, Charlotte, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - PhysiqueMed Clinical Trials, Greensboro, North Carolina
  - Kinston Medical Specialists PA, Kinston, North Carolina
  - Clinical Trials of America, LLC, Mount Airy, North Carolina
  - Trial Management Associates LLC, Wilmington, North Carolina
  - PMG Research of Winston-Salem LLC, Winston-Salem, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Ohio Clinical Research Partners LLC, Akron, Ohio
  - Dr. Deepak Sarwal, MD, Centerville, Ohio
  - UC Health Clinical Trials Office, Cincinnati, Ohio
  - Consultants for Clinical Research Inc., Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Clinical Inquest Center Ltd, Huber Heights, Ohio
  - Springfield Health Care Center, Springfield, Ohio
  - Oklahoma University Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Main Line Gastroenterology, Havertown, Pennsylvania
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania
  - Penn State University Milton S Hershey Medical Center, State College, Pennsylvania
  - ClinSearch LLC, Chattanooga, Tennessee
  - Gastro One, Germantown, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Clinical Research Institute LLC, Arlington, Texas
  - Texas Digestive Disease Consultants - Dallas, Arlington, Texas
  - Texas Digestive Disease Consultants Dallas, Dallas, Texas
  - Texas Digestive Disease Consultants - Southlake, Flower Mound, Texas
  - Gulf Coast Research Group LLC, Houston, Texas
  - The Methodist Hospital Research Institute, Houston, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Houston Endoscopy and Research Center, Houston, Texas
  - Sagact Pllc, San Antonio, Texas
  - San Antonio Military Medical Center, San Antonio, Texas
  - Scott & White Medical Center, Temple, Texas
  - Digestive Health Specialist of Tyler, Tyler, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Vermont, Colchester, Vermont
  - University of Virginia, Charlottesville, Virginia
  - Charlottesville Medical Research Center, Charlottesville, Virginia
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia
  - Emeritas Research Group, Leesburg, Virginia
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - Hunter Holmes Mcguire Ctr, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington
  - University of Washington School of Medicine, Seattle, Washington
  - The Vancouver Clinic, Vancouver, Washington
  - Dean Clinic Oregon, Madison, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (18):
  - Bankstown-Lidcombe Hospital, Bankstown, Australian Capital Territory
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Centre For Digestive Diseases, Five Dock, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Mater Adult Hospital, South Brisbane, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Ballarat Base Hospital, Ballarat
  - Monash Medical Centre Clayton, Bentleigh East
  - St Vincents Hospital Melbourne, Fitzroy
  - Austin Hospital, Heidelberg
  - Royal Brisbane and Women's Hospital, Herston
  - Nepean Hospital, Kingswood, NSW
- Austria (10):
  - LKH Universitaetsklinikum Graz, Graz
  - Medizinische Universitat Innsbruck, Innsbruck
  - Klinikum Klagenfurt am Wörtersee, Klagenfurt
  - KH der Barmherzigen Bruder Linz, Linz
  - a.o.Krankenhaus d.Barmherz.Schwestern Ried, Ried I Innkreis
  - LKH - Universitätsklinikum der PMU Salzburg, Salzburg
  - Ordination Dr. Thomas Haas Darmpraxis Salzburg, Salzburg
  - KH der Barmherzigen Brüder St.Veit an der Glan, Sankt Veit an der Glan
  - Krankenanstalt Rudolfstiftung Wien, Wein
  - AKH Medizinische Universitat Wien, Wein
- Belgium (6):
  - Universitair Ziekenhuis Brussel, Brussels
  - Cliniques Universitaires St Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - UZ Leuven, Leuven
  - CHU Sart Tilman, Liège
  - Centre Hospitalier de Mouscron, Mouscron
- Bulgaria (9):
  - MHAT Sv Nikolay Chudotvorets EOOD, Lom
  - MHAT Kaspela EOOD, Plovdiv
  - MHAT Ruse AD, Rousse
  - Second MHAT Sofia AD, Sofia
  - City Clinic UMHAC EOOD, Sofia
  - UMHAT Sv Ivan Rilski EAD, Sofia
  - UMHAT Tsaritsa Yoanna - ISUL EAD, Sofia
  - Fourth MHAT Sofia EAD, Sofia
  - MHAT Doverie AD, Sofia
- Canada (28):
  - University of Calgary, Calgary, Alberta
  - GI Research Institute, Edmonton, Alberta
  - University of Alberta, Edmonton, Alberta
  - South Edmonton Gastroenterology, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - GI Research Institute, Vancouver, British Columbia
  - PerCuro Clinical Research, Victoria, British Columbia
  - Brandon Medical Arts Clinic, Brandon, Manitoba
  - Barrie GI Associates, Barrie, Ontario
  - McMaster University Health Sciences Center, Hamilton, Ontario
  - London Health Science Center U. Hospital, London, Ontario
  - LHSC Victoria Hospital, London, Ontario
  - Montfort Hospital, Ottawa, Ontario
  - Humber River Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Toronto Liver Centre, Toronto, Ontario
  - Toronto Digestive Disease Associates Inc, Vaughan, Ontario
  - Medicine Professional Corporation, Waterloo, Ontario
  - Tarabain Osman MD, Windsor, Ontario
  - Centre de sante et de services sociaux Champlain Charles Le Moyne, Greenfield Park, Quebec
  - Recherche GCP Research, Montreal, Quebec
  - Hopital Maisonneuve Rosemont dba CIUSSS de lEst de lIle de Montreal, Montreal, Quebec
  - CHUM Hôpital Saint-Luc, Montreal, Quebec
  - McGill University Health Centre Glen Site Royal Victoria Hospital, Montreal, Quebec
  - Recherche Medicale St Jerome Inc, Saint-Jérôme, Quebec
  - CHUS Hopital Fleurimont, Sherbrooke, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan
  - Recherche Clinique Sigma Inc, Québec
- Croatia (6):
  - Clinical Hospital Centre Osijek, Osijek
  - Clinical Hospital Centre Rijeka, Rijeka
  - Clinical Hospital Centre Zagreb, Zagreb
  - Clinical Hospital Dubrava, Zagreb
  - Clinical Hospital Merkur, Zagreb
  - Clinical Hospital Sveti Duh, Zagreb
- Czechia (9):
  - Fakultni nemocnice u sv Anny v Brne, Brno
  - Hepato-Gastroenterologie HK, Hradec Králové
  - Soukroma Gastroenterologicka ambulance a endoskopie, Most
  - PreventaMed, Olomouc
  - CCBR Czech as, Pardubice
  - CCBR Prague CZ, Prague
  - IBD Centrum ISCARE IVF as, Prague
  - Krajska zdravotni, a.s. - Masarykova nemocnice v Usti nad La, Ústí nad Labem
  - Nemocnice Znojmo, Znojmo
- Denmark (7):
  - Aarhus Universitetshospital, Aahus C
  - Alborg University Hospital, Aalborg
  - Nordsjaellands Hospital Frederikssund, Frederikssund
  - Herlev Hospital, Herlev
  - Hvidovre Hospital, Hvidovre
  - Koge Sygehus, Køge
  - Regionshospitalet Silkeborg, Silkeborg
- Estonia (2):
  - West Tallinn Central Hospital, Tallinn
  - Tartu University Hospital, Tartu
- Finland (2):
  - Tampereen yliopistollinen sairaala, Tampere
  - Turunmaan sairaala, Turku
- France (23):
  - CHU Amiens Hopital Sud, Amiens
  - CHU Besancon Hopital Jean Minjoz, Besançon
  - CHU Tours Hopital Trousseau, Chambray-lès-Tours
  - CHU Clermont Ferrand, Clermont-Ferrand
  - Hopital Beaujon, Clichy
  - CHU Dijon - Hopital Bocage Central, Dijon
  - CHU de Grenoble Hopital Nord, Grenoble
  - Groupement Hospitalier Sud Hopital Bicetre, Le Kremlin-Bicêtre
  - Hopital Claude Huriez CHRU Lille, Lille
  - Hopital Nord, Marseille
  - CHU Nantes Hotel Dieu, Nantes
  - CHU Nice Hopital de lArchet 2, Nice
  - Hopital Saint Antoine, Paris
  - Hopital Saint Louis, Paris
  - Groupe Hospitalier Sud Hopital Haut Leveque USN, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU Reims Hopital Robert Debre, Reims
  - CHU Rennes Hopital Pontchaillou, Rennes
  - CHU de Rouen Hopital Charles Nicolle, Rouen
  - CHU Saint Etienne Hopital Nord, Saint-Etienne
  - CHU Strasbourg Hopital Hautepierre, Strasbourg
  - CHU de Toulouse Hopital Rangueil, Toulouse
  - Hopital de Brabois Adultes, Vandœuvre-lès-Nancy
- Germany (35):
  - Charite Universitaetsmedizin Berlin Campus Benjamin Franklin, Berlin
  - Charite Campus Virchow Klinikum, Berlin
  - DRK Kliniken Berlin Westend, Berlin
  - Krankenhaus Waldfriede e V, Berlin
  - Berufsgenossenschaftliches Universitaetsklinikum Bergmannsheil GmbH, Bochum
  - Staedisches Klinikum Brandenburg, Brandenburg
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Dresden
  - Zentrum fuer HIV und Hepatogastroenterologie GmbH, Düsseldorf
  - Universitaetsklinikum Erlangen, Erlangen
  - Kliniken Essen-Mitte, Essen
  - Katholische Kliniken Ruhrhalbinsel GmbH, Essen
  - Agaplesion Markus Krankenhaus, Frankfurt
  - Crohn Colitis Centrum Rhein Main, Frankfurt
  - Universitaetsklinikum FreiburgInnere Med.1, Haematologie, Freiburg im Breisgau
  - Universitaetsklinikum Halle Saale, Halle
  - Asklepios Klinik Hamburg, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitatsklinikum Heidelberg, Heidelberg
  - Praxis fuer Gastroenterologie Dr Ehehal Dr Helmstaedter, Heidelberg
  - Universitaetsklinikum Jena, Jena
  - Universitaetsklinikum Schleswig Holstein Campus Kiel, Kiel
  - University Leipzig, Leipzig
  - Internistische Gemeinschaftspraxis f. Verdauungs- und Stoffwechselerkrankungen, Leipzig
  - EUGASTRO GmbH, Leipzig
  - Medizinisches Zentrum Klinikum Lueneburg, Lüneburg
  - Universitaetsklinikum Magdeburg A oeR, Magdeburg
  - Klinikum Mannheim GmbH Universitaetsklinikum, Mannheim
  - Gastroenterologische Praxis Minden, Minden
  - Isar Klinik GmbH, München
  - Klinikum der Universitaet Muenchen, München
  - Universitaetsklinikum Muenster, Münster
  - Gastro Campus Research, Münster
  - Staedtisches Klinikum Braunschweig gGmbH Standort Salzdahlumer, Niedersachsen
  - Universitaetsklinikum Regensburg, Regensburg
  - Universitaetsklinikum Ulm, Ulm
- Greece (10):
  - University General Hospital of Alexandroupolis, Alexandroupoli
  - General Hospital of Athens Evangelismos, Athens
  - Athens Medical Center, Athens
  - General Hospital of Nikaea Piraeus Ag. Panteleimon, Athens
  - University General Hospital of Heraklion, Heraklion
  - General Hospital of Heraklion Benizeleio Pananeio, Heraklion
  - University General Hospital of Ioannina, Ioannina
  - University General Hospital of Patras, Rio Patras
  - Anticancer Hospital of Thessaloniki THEAGENIO, Thessaloniki
  - General Hospital of Thessaloniki Hippokration, Thessaloniki
- Hungary (18):
  - DRC Gyogyszervizsgalo Kozpont Kft, Balatonfüred
  - Clinexpert Egeszsegugyi Szolg es Ker Kft, Budapest
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
  - Semmelweis Egyetem AOK, Budapest
  - Szent Janos Korhaz es Eszak-budai Egyesitett Korhazak, Budapest
  - Pannonia Maganorvosi Centrum, Budapest
  - Endomedix Diagnosztikai Kozpont, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Szent Pantaleon Korhaz Rendelointezet Dunaujvaros, Dunaújváros
  - Markhot Ferenc Oktato Korhaz es Rendelointezet, Eger
  - Petz Aladar Megyei Oktato Korhaz, Győr
  - Bekes Megyei Pandy Kalman Korhaz, Gyula
  - Somogy Megyei Kaposi Mor Oktato Korhaz, Kaposvár
  - Mohacsi Korhaz, Mohács
  - SzSzB Megyei Korhazak es Egyetemi Oktatokorhaz, Nyíregyháza
  - Mazso-Pharma Kutatas-fejlesztesi Kft, Szeged
  - Clinfan Szolgaltato Kft, Szekszárd
  - Fejer Megyei Szent Gyorgy Egyetemi Oktato Korhaz, Székesfehérvár
- Israel (11):
  - HaEmek Medical Center, Afula
  - Soroka University Medical Center, Beersheba
  - Rambam Health Care Campus, Haifa
  - Wolfson Medical Center, Holon
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah University Hospital, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky Medical Center Department of Hematology, Tel Aviv
  - Assaf Harofeh Medical Center, Ẕerifin
- Italy (20):
  - Azienda Ospedaliero Universitaria Consorziale Policlinico di Bari, Bari
  - Azienda Ospedaliera Universitaria Policlinico Sant Orsola Malpighi, Bologna
  - Azienda Ospedaliera Universitaria Policlinico G Martino, Messina
  - Fondazione IRCCS CA Granda Ospedale Maggiore Policlinico, Milan
  - Seconda Universita Degli Studi Di Napoli, Naples
  - Azienda Ospedaliera Universitaria Federico II, Napoli, Campania
  - Hospital of Di Padova, Padua
  - Azienda Ospedaliera Vincenzo Cervello, Palermo
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Universita Campus Bio-Medico di Roma, Roma
  - Ospedale Sandro Pertini, Roma
  - Complesso Integrato Columbus, Roma
  - Policlinico Universitario Agostino Gemelli, Roma
  - Azienda Ospedaliera San Camillo Forlanini, Rome
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata, Rome
  - Istituto Clinico Humanitas, Rozzano (MI)
  - Azienda Ospedaliera Universitaria OO. RR. S. Giovanni di Dio e Ruggi dAragona, Salerno
  - IRCCS Policlinico San Donato, San Donato Milanese
  - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo FG
- Latvia (3):
  - Digestive Diseases Center Gastro, Riga
  - Riga East Clinical University Hospital clinic Gailezers, Riga
  - Pauls Stradins Clinical University Hospital, Riga
- Malaysia (5):
  - Hospital Sultanah Bahiyah, Alor Star, Kedah
  - Hospital Universiti Sains Malaysia, Kelantan, Kelantan
  - Hospital Raja Perempuan Zainab II, Kota Bharu, Kelantan
  - University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur
  - Hospital Ampang, Ampang, Selangor
- Netherlands (10):
  - VU Medisch Centrum, Amsterdam
  - Academisch Medisch Centrum, Amsterdam
  - Amphia Ziekenhuis, Breda
  - Universitair Medisch Centrum Groningen, Groningen
  - Leiden Universitair Medisch Centrum, Leiden
  - Medisch Centrum Haaglanden,Antoniushoeve, Leidschendam
  - Radboudumc, Nijmegen
  - Zuyderland Medisch Centrum, Sittard-Geleen
  - St. Elisabeth Ziekenhuis, Tilburg
  - University Medical Center Utrecht, Utrecht
- Waikato Hospital, Hamilton, New Zealand
- Norway (5):
  - Sykehuset Ostfold Fredrikstad, Fredrikstad
  - Akershus universitetssykehus HF, Lørenskog
  - Oslo Universitetssykehus HF Ulleval, Oslo
  - Oslo Universitetssykehus Rikshospitalet, Oslo
  - Stavanger Unviversitetssjukehus Helse Stavanger HF, Stavanger
- Poland (16):
  - SP ZOZ Wojewodzki Szpital Zespolony im. J. Sniadeckiego, Bialystok
  - Clinsante S.C. Osrodek Badan Klinicznych, Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Niepubliczny Zaklad Opieki Zdrowotnej POLIMEDICA, Kielce
  - Indywidualna Praktyka Lekarska Maciej Zymla, Knurów
  - Centrum Medyczne Plejady, Krakow
  - LUX MED Sp. z o.o., Krakow
  - SPZOZ Szpital Uniwersytecki w Krakowie, Krakow
  - SPZOZ Uniwersytecki Szpital Kliniczny im. Wojskowej Akademii Medycznej - Centralny Szpital Weteranow, Lodz
  - Centrum Medyczne AMED, Lodz
  - GASTROMED Sp.zo.o., Lublin
  - Ai Centrum Medyczne Sp. Z O.O. Sp.K., Poznan
  - Centrum Medyczne Medyk, Rzeszów
  - Endoskopia Sp. z o.o., Sopot
  - Nzoz Vivamed, Warsaw
  - LexMedica Osrodek Badan Klinicznych, Wroclaw
- Portugal (6):
  - Hospital de Braga, Braga
  - Centro Hospitalar E Universitario de Coimbra EPE, Coimbra
  - Hospital da Senhora da Oliveira Guimaraes, Guimarães
  - Hospital Da Luz, Lisbon
  - Centro Hospitalar de Sao Joao, EPE, Porto
  - Centro Hospitalar do Alto Minho - Unidade Local de Saúde do Alto Minho, EPE, Viana do Castelo
- Romania (5):
  - S.C MedLife S.A, Bucharest
  - Tvm Med Serv Srl, Cluj-Napoca
  - Spitalul Clinic Judetean de Urgente Sf. Spiridon, Iași
  - CMI Dr. Tirnaveanu Amelita, Oradea
  - Centrul de Gastroenterologie Dr. Goldis, Timișoara
- Russia (19):
  - Irkutsk State Medical Academy of Continuing Education, Irkutsk
  - TSBIH Territorial Clinical Hospital, Krasnoyarsk
  - Medical Center Stolitsa-Medikl, Moscow
  - SBHI of NN region RCH of NN n.a. N.A.Semashko, Nizhny Novgorod
  - SBEIHPE Novosibirsk State Medical University, Novosibirsk
  - RSHI State Novosibirsk Regional Clinical Hospital, Novosibirsk
  - FSBI Scientific Research Institute of Physyology and Basic Medicine under the SB of RAMS, Novosibirsk
  - BHI of Omsk region Clinical Oncology Dispensary, Omsk
  - SBEI of HPE Omsk State Medical Academy Ministry of healthcare of RF, Omsk
  - SBIH of Perm territory City Clinical Hospital 2 na Fedor Khristoforovich Gral, Perm
  - Evromedservis, Pushkin
  - SEIHPE Rostov State Medical University of MoH of RF, Rostov-on-Don
  - City Mariinskaya Hospital, Saint Petersburg
  - SPb SBIH City Hospital # 26, Saint Petersburg
  - Private Educational Institution of Higher Education Medical university REAVIZ, Samara
  - NonState Healthcare Institution Central Clinical Hospital, Samara station JSC Russian Railways, Samara
  - SHI Regional Clinical Hospital, Saratov
  - SBI of Healthcare of Leningrad region Clinical Interregional Hospital of Tosno, Tosno
  - SBHI of Yaroslavl Region Clinical Hospital 8, Yaroslavl
- Serbia (7):
  - Clinical Center of Serbia, Belgrade
  - Clinical Center Zvezdara, Belgrade
  - Military Medical Academy, Belgrade
  - Clinical Center Bezanijska Kosa, Belgrade
  - Clinical Center Zemun, Belgrade
  - Clinical Center Kragujevac, Kragujevac
  - Clinical Center Nis, Niš
- Slovakia (13):
  - Fakultna nemocnica s poliklinikou F. D. Roosevelta, Banská Bystrica
  - Alian s.r.o., Bardejov
  - Univerzitna nemocnica Bratislava Nemocnica Ruzinov, Bratislava
  - Gastroentero-Hepatologicke centrum THALION, Bratislava
  - Nemocnica A.Lena Humenne n o, Humenné
  - B & B MED, s.r.o., Košice
  - KARDIO 1 s.r.o., Lučenec
  - Gastroeneterologicka ambulancia MUDr. Peter Hegyi s.r.o., Malacky
  - Fakultna nemocnica Nitra, Nitra
  - KM Management, spol. s r.o., Nitra
  - GASTRO I., s.r.o., Prešov
  - Nemocnica s poliklinikou sv Barbory Roznava a s, Rožňava
  - Fakultna nemocnica s poliklinikou Zilina, Žilina
- South Korea (14):
  - Dong-A University Hospital, Busan
  - Pusan National University Hospital, Busan
  - Yeungnam University Medical Center, Daegu
  - Hanyang Univerisy Guri Hospital, Guri-si
  - CHA Bundang Medical Center CHA University, Seongnam-si
  - Seoul National University Bundang Hospital, Seongnam-si
  - Kyung Hee University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Asan Medical Center, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - The Catholic University of Korea, St.Vicent's Hospital, Suwon
- Spain (12):
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital del Mar, Barcelona
  - Hospital Clinic I Provincial de Barcelona, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario de la Princesa, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
  - Corporacion Sanitaria Parc Tauli, Sabadell
  - Hospital Universitario Infanta Sofia, San Sebastián de los Reyes
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Miguel Servet, Zaragoza
- Sweden (3):
  - Sodersjukhuset, Stockholm
  - Danderyds Sjukhus AB, Stockholm
  - Akademiska Sjukhuset, Uppsala
- Switzerland (5):
  - Universitaetsspital Basel, Basel
  - Inselspital - Universitaetsspital Bern, Bern
  - Crohn-Colitis Zentrum Bern Gemeinschaftspraxis Balsiger Seibold und Partner, Bern
  - Kantonsspital St.Gallen, Sankt Gallen
  - Universitaetsspital Zuerich, Zurich
- Turkey (Türkiye) (16):
  - Ankara University Medical Faculty, Ankara
  - Hacettepe University Medical Faculty, Ankara
  - Turkiye Yuksek Ihtisas Hospital, Ankara
  - Gazi University Medical Faculty, Ankara
  - Firat University Medical Faculty, Elâzığ
  - Gaziantep University Medical Faculty Sahinbey Educational Research Hospital, Gaziantep
  - Yeditepe University Medical School Hospital, Istanbul
  - Istanbul University Cerrahpasa Medical Faculty Hospital, Istanbul
  - Acibadem Fulya Hospital, Istanbul
  - Haydarpasa Numune Training and Research Hospital, Istanbul
  - Istanbul Medeniyet Uni Goztepe Training&Res Hosp, Istanbul
  - Marmara University Pendik Training and Research Hospital, Istanbul
  - Ege University Medical Faculty, Izmir
  - Inonu Uni. Med. Fac., Malatya
  - Mersin University Medical Faculty, Mersin
  - Kocaeli Derince Training and Research Hospital, Umuttepe Kocaeli
- Ukraine (18):
  - RCI Chernivtsi Regional Clinical Hospital Dept of Surgery Bukovinian SMU, Chernivtsi
  - CI of PH Kharkiv CCH #2, Kharkiv
  - GI L.T.Malaya Therapy National Institute of the NAMS of Ukraine, Kharkiv
  - Treatment-Diagnostic Center of Private Enterprise of PMF Atsynus, Kirovohrad
  - Ukrainian-German Antiulcer Gastroenterological Center BYK-Kyiv LLC, Kyiv
  - Kyiv City Clinical Hospital #1, Kyiv
  - SI Republican Clinical Hospital of the MOHU Dept of Gastroenterology O.O.Bogomolets NMU, Kyiv
  - Lviv Regional Clinical Hospital D Halytskyi Lviv NMU, Lviv
  - Lviv Municipal City Clinical Hospital #5 Dept of Therapy D.Halytsky Lviv NMU, Lviv
  - CI Odesa Regional Clinical Hospital, Odesa
  - Communal Institution City Policlinic #20 Cabinet of Gastroenterology, Odesa
  - M.V. Sklifosovskyi Poltava RCH Outpatient UMSA HSEIU Ukrainian Medical Stomatological Academy, Poltava
  - CI of SRC Sumy RCH Dept of Rheumatology Sumy SU MI, Sumy
  - Ternopil City Communal Emergency Medical Care Hospital, Ternopil
  - M.I. Pyrogov VRCH Dept of Gastroenterology M.I. Pyrogov VNMU, Vinnytsia
  - SRI of Invalid Rehabilitation EST Complex of Vinnytsia M.I.Pyrogov NMU MOHU, Vinnytsia
  - SI Branch CH of Zaporizhzhia Station-2 of SE Prydniprovska Railway Dept of Surgery Zaporizhzhia SMU, Zaporizhia
  - CI Zaporizhzhia Regional Clinical Hospital of ZRC, Zaporizhzhya
- United Kingdom (15):
  - Queen Elizabeth Hospital, Birmingham
  - Bristol Royal Infirmary, Bristol
  - Royal Devon and Exeter Hospital Wonford, Exeter
  - Queen Elizabeth University Hospital, Glasgow
  - Glasgow Royal Infirmary, Glasgow, Scotland
  - Hull Royal Infirmary, Hull
  - Royal London Hospital, London
  - St Marys Hospital, London
  - Manchester Royal Infirmary, Manchester
  - University Hospital of South Manchester NHS Foundation Trust -Wythenshawe Hospital - North West Lung, Manchester
  - Nottingham University Hospitals Queens Medical Centre, Nottingham
  - John Radcliffe Hospital, Oxford
  - Borders General Hospital, Roxburghshire
  - Royal Shrewsbury Hospital, Shrewsbury
  - Southampton General Hospital, Southhampton

REFERENCES:
- [Background] Gold SL, Cohen-Mekelburg S, Schneider Y, Steinlauf A. Perianal Fistulas in Patients With Crohn's Disease, Part 2: Surgical, Endoscopic, and Future Therapies. Gastroenterol Hepatol (N Y). 2018 Sep;14(9):521-528. PMID 30364296
- [Derived] Sands BE, Feagan BG, Sandborn WJ, Schreiber S, Peyrin-Biroulet L, Frederic Colombel J, Rossiter G, Usiskin K, Ather S, Zhan X, D'Haens G. Mongersen (GED-0301) for Active Crohn's Disease: Results of a Phase 3 Study. Am J Gastroenterol. 2020 May;115(5):738-745. doi: 10.14309/ajg.0000000000000493. PMID 31850931

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study centers within the United States and Canada, Australia, Eastern and Western Europe, Korea and Russia.
Pre-assignment Details: Treatment assignment at baseline (Week 0) was stratified based on concomitant use of corticosteroids (yes/no), concomitant use of immunosuppressants (yes/no) or and previous exposure to biologics (yes/no),
Groups:
- Placebo: Participants received placebo daily up to week 52.
- GED-0301 160 mg / GED-0301 40 mg 4 Week Alt: Participants received GED-0301 160 mg daily for 12 weeks, followed by alternating placebo daily for 4 weeks and GED-0301 40 mg daily for 4 weeks, up to week 52.
- GED-0301 160 mg / GED-0301 40 mg: Participants received GED-0301 160 mg daily for 12 weeks, followed by continuous GED-0301 40 mg daily, up to week 52.
- GED-0301 160 mg / GED-0301 160 mg 4 Week Alt: Participants received GED-0301 160 mg daily for 12 weeks, followed by alternating placebo daily for 4 weeks and GED-0301 160 mg daily for 4 weeks, up to week 52.
Period: Overall Double-Blind Period Weeks 0-52
Arm/Group | Placebo | GED-0301 160 mg / GED-0301 40 mg 4 Week Alt | GED-0301 160 mg / GED-0301 40 mg | GED-0301 160 mg / GED-0301 160 mg 4 Week Alt
Started | 174 | 176 | 176 | 175
Completed | 10 | 8 | 14 | 9
Not Completed | 164 | 168 | 162 | 166
Not completed — Study Terminated by Sponsor | 61 | 56 | 48 | 58
Not completed — Adverse Event | 11 | 15 | 15 | 12
Not completed — Pregnancy | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 15 | 14 | 14 | 13
Not completed — Withdrawal by Subject | 10 | 4 | 13 | 5
Not completed — Miscellaneous | 1 | 2 | 0 | 2
Not completed — Lost to Follow-up | 0 | 1 | 1 | 1
Not completed — Non-Compliance with Study Drug | 0 | 0 | 1 | 2
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 2
Not completed — Early Escape | 66 | 76 | 69 | 70
Period: Follow-Up Period Weeks 0 to 52
Arm/Group | Placebo | GED-0301 160 mg / GED-0301 40 mg 4 Week Alt | GED-0301 160 mg / GED-0301 40 mg | GED-0301 160 mg / GED-0301 160 mg 4 Week Alt
Started | 57 | 51 | 56 | 47
Completed | 57 | 51 | 56 | 47
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) population consisted of all participants who were randomized and received at least 1 dose of investigational product (IP). Treatment assignment at Week 0 visit was based on concomitant use of corticosteroids (yes/no), concomitant use of immunosuppressants (yes/no) or and previous exposure to biologics (yes/no),
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | GED-0301 160 mg / GED-0301 40 mg 4 Week Alt | GED-0301 160 mg / GED-0301 40 mg | GED-0301 160 mg / GED-0301 160 mg 4 Week Alt | Total
Number analyzed (Participants) | 174 | 176 | 176 | 175 | 701
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.5 (12.88) | 37.6 (12.84) | 39.6 (12.90) | 38.2 (12.47) | 38.5 (12.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 98 | 92 | 80 | 346
  Male | 98 | 78 | 84 | 95 | 355
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 0 | 2
  Asian | 11 | 2 | 8 | 8 | 29
  Black or African American | 4 | 4 | 2 | 2 | 12
  White | 150 | 165 | 152 | 158 | 625
  Not Collected or Reported | 5 | 4 | 9 | 5 | 23
  Other (No classification) | 3 | 1 | 4 | 2 | 10
Duration of Crohn's Disease [Mean (Standard Deviation); unit: Years] | 9.57 (9.106) | 8.63 (7.877) | 9.84 (8.746) | 10.15 (9.353) | 9.54 (8.786)
Baseline Crohn's Disease Activity (CDAI) Score [Mean (Standard Deviation); unit: Units on a Scale] — The Crohn's Disease Activity Index (CDAI) is used to quantify the signs and symptoms of Crohn's disease and the effect on patient's quality of life. It consists of 8 variables which include patient reported outcomes over a 7 day period and physician assessments which are scored numerically and weighted. Scores range from 0 to 600, with the most severe disease defined >450. Population: 1 participant CDAI was missing in the placebo arm and the GED-0301 160 mg/ 40 mg 4 Week Alt arm.
  Units on a Scale
    number analyzed (Participants) | 173 | 175 | 176 | 175 | 699
    (all) | 307.9 (64.31) | 292.8 (69.33) | 308.3 (65.50) | 309.9 (66.32) | 304.7 (66.61)
Baseline Endoscopic Score for Crohn's Disease (Central Read) [Mean (Standard Deviation); unit: Units on a Scale] — The Simple Endoscopic Score for Crohn's Disease (SES-CD) is a validated index used to quantify the presence and size of ulcers, extent of ulcerated surface, extent of affected surface and presence and type of narrowings across 5 segments across the distal ileum and colon. Scores range from 0 to 60 with higher scores reflecting more severe disease. Population: 1 participant endoscopic was missing in the placebo arm.
  Units on a Scale
    number analyzed (Participants) | 173 | 176 | 176 | 175 | 700
    (all) | 14.4 (7.88) | 14.3 (8.41) | 13.8 (7.69) | 14.5 (8.30) | 14.2 (8.06)

OUTCOME MEASURES:

1. Secondary Outcome: Percentage of Participants Who Achieved Clinical Remission at Week 52
Description: Clinical remission is defined as a CDAI score < 150 and is used to quantify the signs and symptoms of Crohn's disease and the effect on patient's quality of life. It consists of 8 variables which include patient reported outcomes over a 7 day period and physician assessments which are scored numerically and weighted. Scores range from 0 to 600, with the most severe disease defined >450.
Time Frame: Week 52
Population: ITT population; Includes participants who had either completed that timepoint visit or discontinued at any time due to reasons other than study terminated by sponsor. NRI.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | GED-0301 160 mg / GED-0301 40 mg 4 Week Alt | GED-0301 160 mg / GED-0301 40 mg | GED-0301 160 mg / GED-0301 160 mg 4 Week Alt
Number analyzed (Participants) | 113 | 120 | 128 | 117
percentage of participants | 5.3 [2.5 to 11.1] | 2.5 [0.9 to 7.1] | 9.4 [5.4 to 15.7] | 3.4 [1.3 to 8.5]
Statistical Analysis 1: Comparison: Placebo vs GED-0301 160 mg / GED-0301 40 mg 4 Week Alt; Test type: Superiority; p = 0.2523, Cochran-Mantel-Haenszel; Stratified Difference = -2.9, 95% CI 2-sided [-9.7 to 3.9] — The weighted average of the treatment differences across the strata with the CMH weights
Statistical Analysis 2: Comparison: Placebo vs GED-0301 160 mg / GED-0301 40 mg; Test type: Superiority; p = 0.1626, Cochran-Mantel-Haenszel; Slope = 4.8, 95% CI 2-sided [-3.0 to 11.8] — The weighted average of the treatment differences across the strata with the CMH weights
Statistical Analysis 3: Comparison: Placebo vs GED-0301 160 mg / GED-0301 160 mg 4 Week Alt; Test type: Superiority; p = 0.4420, Cochran-Mantel-Haenszel; Stratified Difference = -2.1, 95% CI 2-sided [-9.1 to 5.3] — The weighted average of the treatment differences across the strata with the CMH weights

2. Secondary Outcome: Percentage of Participants With Endoscopic Response-50 Centrally Read at Week 52
Description: An endoscopic response-50 is defined as a reduction of at least 50% compared with baseline in simple endoscopic score for Crohn's Disease (SES-CD). The SES-CD assesses the size of mucosal ulcers, the extent of ulcerated surface, the extent of affected surface, and the presence and type of narrowings. Scores range from 0 to 60 with higher scores reflecting more severe disease. The SES-CD calculations include:
  * Ulcers scored as:
    0: no
    1. aphthous (0.1-0.5 cm)
    2. large (0.5-2 cm)
    3. very large (>2 cm)
  * Surface involved disease 0: 0%
    1. <50%
    2. 50-75%
    3. >75%
  Surface involved by ulcerations:
  0: 0%
  1. <10%
  2. 10-30%
  3. >30% - Narrowings:
  0: No
  1. Single, can be passed
  2. Multiple, can be passed
  3. Cannot be passed Grand Total = SES-CD score
Time Frame: Week 52
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | GED-0301 160 mg / GED-0301 40 mg 4 Week Alt | GED-0301 160 mg / GED-0301 40 mg | GED-0301 160 mg / GED-0301 160 mg 4 Week Alt
Number analyzed (Participants) | 113 | 120 | 128 | 117
percentage of participants | 3.5 [1.4 to 8.7] | 0.8 [0.1 to 4.6] | 1.6 [0.4 to 5.5] | 1.7 [0.5 to 6.0]
Statistical Analysis 1: Comparison: Placebo vs GED-0301 160 mg / GED-0301 40 mg 4 Week Alt; Test type: Superiority; p = 0.1799, Cochran-Mantel-Haenszel; Stratified Difference = -2.6, 95% CI 2-sided [-9.5 to 5.0] — The weighted average of the treatment differences across the strata with the CMH weights
Statistical Analysis 2: Comparison: Placebo vs GED-0301 160 mg / GED-0301 40 mg; Test type: Superiority; p = 0.2309, Cochran-Mantel-Haenszel; Stratified Difference = -2.4, 95% CI 2-sided [-9.4 to 4.9] — The weighted average of the treatment differences across the strata with the CMH weights
Statistical Analysis 3: Comparison: Placebo vs GED-0301 160 mg / GED-0301 160 mg 4 Week Alt; Test type: Superiority; p = 0.3264, Cochran-Mantel-Haenszel; Stratified Difference = -2.1, 95% CI 2-sided [-9.1 to 4.6] — The weighted average of the treatment differences across the strata with the CMH weights

3. Secondary Outcome: The Percentage of Participants Who Achieved a Clinical Response at Week 12
Description: A clinical response is defined as a CDAI score decrease from baseline ≥ 100 points. The CDAI is used to quantify the signs and symptoms of Crohn's disease and the effect on patient's quality of life. It consists of 8 variables which include patient reported outcomes over a 7 day period and physician assessments which are scored numerically and weighted. Scores range from 0 to 600, with the most severe disease defined >450.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | GED-0301 160 mg / GED-0301 40 mg 4 Week Alt | GED-0301 160 mg / GED-0301 40 mg | GED-0301 160 mg / GED-0301 160 mg 4 Week Alt
Number analyzed (Participants) | 160 | 162 | 164 | 157
percentage of participants | 44.4 [36.9 to 52.1] | 32.1 [25.4 to 39.6] | 34.1 [27.3 to 41.7] | 33.8 [26.8 to 41.5]
Statistical Analysis 1: Comparison: Placebo vs GED-0301 160 mg / GED-0301 40 mg 4 Week Alt; Test type: Superiority; p = 0.0299, Cochran-Mantel-Haenszel; Stratified Difference = -11.7, 95% CI 2-sided [-22.0 to -1.1] — The weighted average of the treatment differences across the strata with the CMH weights
Statistical Analysis 2: Comparison: Placebo vs GED-0301 160 mg / GED-0301 40 mg; Test type: Superiority; p = 0.0582, Cochran-Mantel-Haenszel; Stratified difference = -9.9, 95% CI 2-sided [-20.3 to 0.7] — The weighted average of the treatment differences across the strata with the CMH weights
Statistical Analysis 3: Comparison: Placebo vs GED-0301 160 mg / GED-0301 160 mg 4 Week Alt; Test type: Superiority; p = 0.0741, Cochran-Mantel-Haenszel; Stratified difference = -9.7, 95% CI 2-sided [-20.1 to 1.0] — The weighted average of the treatment differences across the strata with the Cochran-Mantel-Haenszel (CMH) weights

4. Secondary Outcome: The Percentage of Participants Who Achieved a Clinical Response at Week 4
Description: A clinical response is defined as a decrease from baseline in CDAI ≥ 100 points. The Crohn's Disease Activity Index is used to quantify the signs and symptoms of Crohn's disease and the effect on patient's quality of life. It consists of 8 variables which include patient reported outcomes over a 7 day period and physician assessments which are scored numerically and weighted. Scores range from 0 to 600, with the most severe disease defined >450.
Time Frame: Week 4
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | GED-0301 160 mg / GED-0301 40 mg 4 Week Alt | GED-0301 160 mg / GED-0301 40 mg | GED-0301 160 mg / GED-0301 160 mg 4 Week Alt
Number analyzed (Participants) | 169 | 172 | 170 | 169
percentage of participants | 34.3 [27.6 to 41.8] | 28.5 [22.3 to 35.6] | 32.4 [25.8 to 39.7] | 27.8 [21.6 to 35.0]
Statistical Analysis 1: Comparison: Placebo vs GED-0301 160 mg / GED-0301 40 mg 4 Week Alt; Test type: Superiority; p = 0.2493, Cochran-Mantel-Haenszel; Stratified difference = -5.8, 95% CI 2-sided [-15.5 to 4.0] — The weighted average of the treatment differences across the strata with the Cochran-Mantel-Haenszel (CMH) weights
Statistical Analysis 2: Comparison: Placebo vs GED-0301 160 mg / GED-0301 40 mg; Test type: Superiority; p = 0.7160, Cochran-Mantel-Haenszel; Stratified difference = -1.8, 95% CI 2-sided [-11.8 to 8.2] — The weighted average of the treatment differences across the strata with the Cochran-Mantel-Haenszel (CMH) weights
Statistical Analysis 3: Comparison: Placebo vs GED-0301 160 mg / GED-0301 160 mg 4 Week Alt; Test type: Superiority; p = 0.2452, Cochran-Mantel-Haenszel; Stratified difference = -5.8, 95% CI 2-sided [-15.5 to 4.1] — The weighted average of the treatment differences across the strata with the Cochran-Mantel-Haenszel (CMH) weights

5. Secondary Outcome: The Percentage of Participants Who Achieved a Clinical Remission at Week 4
Description: A clinical remission is a CDAI score < 150. The Crohn's Disease Activity Index is used to quantify the signs and symptoms of Crohn's disease and the effect on patient's quality of life. It consists of 8 variables which include patient reported outcomes over a 7 day period and physician assessments which are scored numerically and weighted. Scores range from 0 to 600, with the most severe disease defined >450.
Time Frame: Week 4
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | GED-0301 160 mg / GED-0301 40 mg 4 Week Alt | GED-0301 160 mg / GED-0301 40 mg | GED-0301 160 mg / GED-0301 160 mg 4 Week Alt
Number analyzed (Participants) | 169 | 172 | 170 | 169
percentage of participants | 20.1 [14.8 to 26.8] | 18.6 [13.5 to 25.1] | 16.5 [11.6 to 22.8] | 15.4 [10.7 to 21.6]
Statistical Analysis 1: Comparison: Placebo vs GED-0301 160 mg / GED-0301 40 mg 4 Week Alt; Test type: Superiority; p = 0.7541, Cochran-Mantel-Haenszel; Stratified difference = -1.3, 95% CI 2-sided [-9.8 to 7.1] — The weighted average of the treatment differences across the strata with the Cochran-Mantel-Haenszel (CMH) weights
Statistical Analysis 2: Comparison: Placebo vs GED-0301 160 mg / GED-0301 40 mg; Test type: Superiority; p = 0.3784, Cochran-Mantel-Haenszel; Stratified difference = -3.7, 95% CI 2-sided [-12.0 to 4.6] — The weighted average of the treatment differences across the strata with the Cochran-Mantel-Haenszel (CMH) weights
Statistical Analysis 3: Comparison: Placebo vs GED-0301 160 mg / GED-0301 160 mg 4 Week Alt; Test type: Superiority; p = 0.2865, Cochran-Mantel-Haenszel; Stratified difference = -4.4, 95% CI 2-sided [-12.6 to 3.8] — The weighted average of the treatment differences across the strata with the Cochran-Mantel-Haenszel (CMH) weights

6. Secondary Outcome: The Percentage of Participants Who Achieved a Corticosteroid-Free Clinical Remission at Week 52
Description: The percentage of participants who were receiving oral corticosteroids for Crohn's disease, at baseline and achieved a clinical remission (CDAI score <150) at Week 52 without corticosteroids. The Crohn's Disease Activity Index is used to quantify the signs and symptoms of Crohn's disease and the effect on patient's quality of life. It consists of 8 variables which include patient reported outcomes over a 7 day period and physician assessments which are scored numerically and weighted. Scores range from 0 to 600, with the most severe disease defined >450.
Time Frame: Week 52
Population: ITT population; includes participants who received oral corticosteroids at baseline and had either completed that timepoint visit or discontinued at any time due to reasons other than study terminated by sponsor. NRI.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | GED-0301 160 mg / GED-0301 40 mg 4 Week Alt | GED-0301 160 mg / GED-0301 40 mg | GED-0301 160 mg / GED-0301 160 mg 4 Week Alt
Number analyzed (Participants) | 46 | 39 | 43 | 42
percentage of participants | 2.2 [0.4 to 11.3] | 0.0 [0.0 to 9.0] | 7.0 [2.4 to 18.6] | 2.4 [0.4 to 12.3]
Statistical Analysis 1: Comparison: Placebo vs GED-0301 160 mg / GED-0301 40 mg 4 Week Alt; 2-sided 95% CI were based on the unstratified Newcombe method; Test type: Superiority; p = 0.3572, Cochran-Mantel-Haenszel; p-values were based on the unstratified CMH test when 1 and only 1 of the 2 treatment groups being compared had no subjects in a stratum; Unstratified CMH = -2.2, 95% CI 2-sided [-11.3 to 7.0] — The weighted average of the treatment differences across the strata with the CMH weights
Statistical Analysis 2: Comparison: Placebo vs GED-0301 160 mg / GED-0301 40 mg; Test type: Superiority; p = 0.2823, Cochran-Mantel-Haenszel; Stratified difference = 4.7, 95% CI 2-sided [-8.8 to 18.9] — The weighted average of the treatment differences across the strata with the CMH weights
Statistical Analysis 3: Comparison: Placebo vs GED-0301 160 mg / GED-0301 160 mg 4 Week Alt; Test type: Superiority; p > 0.9999, Cochran-Mantel-Haenszel; Stratified difference = 0.0, 95% CI 2-sided [-12.8 to 13.7] — The weighted average of the treatment differences across the strata with the CMH weights

7. Secondary Outcome: Percentage of Participants Who Achieved a Sustained Clinical Remission at Both Week 12 and 52
Description: For participants who achieved a sustained clinical remission at both week 12 and 52, the clinical remission is a CDAI score < 150. The Crohn's Disease Activity Index is used to quantify the signs and symptoms of Crohn's disease and the effect on patient's quality of life. It consists of 8 variables which include patient reported outcomes over a 7 day period and physician assessments which are scored numerically and weighted. Scores range from 0 to 600, with the most severe disease defined >450.
Time Frame: Weeks 12 and 52
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | GED-0301 160 mg / GED-0301 40 mg 4 Week Alt | GED-0301 160 mg / GED-0301 40 mg | GED-0301 160 mg / GED-0301 160 mg 4 Week Alt
Number analyzed (Participants) | 113 | 120 | 128 | 117
percentage of participants | 2.7 [0.9 to 7.5] | 2.5 [0.9 to 7.1] | 3.9 [1.7 to 8.8] | 1.7 [0.5 to 5.0]
Statistical Analysis 1: Comparison: Placebo vs GED-0301 160 mg / GED-0301 40 mg 4 Week Alt; Test type: Superiority; p = 0.8031, Cochran-Mantel-Haenszel; Stratified difference = -0.5, 95% CI 2-sided [-6.7 to 5.9] — The weighted average of the treatment differences across the strata with the CMH weights
Statistical Analysis 2: Comparison: Placebo vs GED-0301 160 mg / GED-0301 40 mg; Test type: Superiority; p = 0.5583, Cochran-Mantel-Haenszel; Stratified difference = 1.4, 95% CI 2-sided [-5.1 to 7.3] — The weighted average of the treatment differences across the strata with the CMH weights
Statistical Analysis 3: Comparison: Placebo vs GED-0301 160 mg / GED-0301 160 mg 4 Week Alt; Test type: Superiority; p = 0.6123, Cochran-Mantel-Haenszel; Stratified difference = -1.0, 95% CI 2-sided [-7.2 to 6.8]; The weighted average of the treatment differences across the strata with the CMH weights

8. Secondary Outcome: Percentage of Participants With Endoscopic Response-25 Centrally Read at Week 12
Description: An endoscopic response-25 is defined as a reduction of at least 25% compared with baseline in simple endoscopic score for Crohn's disease (SES-CD). The SES-CD assesses the size of mucosal ulcers, the extent of ulcerated surface, the extent of affected surface, and the presence and type of narrowings. Scores range from 0 to 60 with higher scores reflecting more severe disease. The SES-CD calculations include:
  * Ulcers scored as:
    0: no
    1. aphthous (0.1-0.5 cm)
    2. large (0.5-2 cm)
    3. very large (>2 cm)
  * Surface involved disease 0: 0%
    1. <50%
    2. 50-75%
    3. >75%
  Surface involved by ulcerations:
  0: 0%
  1. <10%
  2. 10-30%
  3. >30% - Narrowings:
  0: No
  1. Single, can be passed
  2. Multiple, can be passed
  3. Cannot be passed Grand Total = SES-CD score
Time Frame: Week 0, Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | GED-0301 160 mg / GED-0301 40 mg 4 Week Alt | GED-0301 160 mg / GED-0301 40 mg | GED-0301 160 mg / GED-0301 160 mg 4 Week Alt
Number analyzed (Participants) | 160 | 162 | 164 | 157
percentage of participants | 28.1 [21.7 to 35.5] | 17.3 [12.2 to 23.8] | 27.4 [21.2 to 34.7] | 24.2 [18.2 to 31.5]
Statistical Analysis 1: Comparison: Placebo vs GED-0301 160 mg / GED-0301 40 mg 4 Week Alt; Test type: Superiority; p = 0.0239, Cochran-Mantel-Haenszel; Stratified difference = -10.6, 95% CI 2-sided [-19.6 to -1.4] — The weighted average of the treatment differences across the strata with the CMH weights
Statistical Analysis 2: Comparison: Placebo vs GED-0301 160 mg / GED-0301 40 mg; Test type: Superiority; p = 0.8334, Cochran-Mantel-Haenszel; Stratified difference = -1.0, 95% CI 2-sided [-10.8 to 8.7] — The weighted average of the treatment differences across the strata with the CMH weights
Statistical Analysis 3: Comparison: Placebo vs GED-0301 160 mg / GED-0301 160 mg 4 Week Alt; Test type: Superiority; p = 0.4383, Cochran-Mantel-Haenszel; Stratified difference = -3.9, 95% CI 2-sided [-13.5 to 5.8] — The weighted average of the treatment differences across the strata with the Cochran-Mantel-Haenszel (CMH) weights

9. Secondary Outcome: Percentage of Participants With Endoscopic Remission Centrally Read at Week 52
Description: Endoscopic remission is defined as a simple endoscopic score for Crohn's disease (SES-CD) of ≤2 at the specified timeframe. The SES-CD assesses the size of mucosal ulcers, the extent of ulcerated surface, the extent of affected surface, and the presence and type of narrowings. Scores range from 0 to 60 with higher scores reflecting more severe disease. The SES-CD calculations include:
  * Ulcers scored as:
    0: no
    1. aphthous (0.1-0.5 cm)
    2. large (0.5-2 cm)
    3. very large (>2 cm)
  * Surface involved disease 0: 0%
    1. <50%
    2. 50-75%
    3. >75%
  Surface involved by ulcerations:
  0: 0%
  1. <10%
  2. 10-30%
  3. >30% - Narrowings:
  0: No
  1. Single, can be passed
  2. Multiple, can be passed
  3. Cannot be passed Grand Total = SES-CD score
Time Frame: Week 52
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | GED-0301 160 mg / GED-0301 40 mg 4 Week Alt | GED-0301 160 mg / GED-0301 40 mg | GED-0301 160 mg / GED-0301 160 mg 4 Week Alt
Number analyzed (Participants) | 113 | 120 | 128 | 117
percentage of participants | 2.7 [0.9 to 7.5] | 0.8 [0.1 to 4.6] | 0.8 [0.1 to 4.3] | 0.9 [0.2 to 4.7]
Statistical Analysis 1: Comparison: Placebo vs GED-0301 160 mg / GED-0301 40 mg 4 Week Alt; Test type: Superiority; p = 0.3573, Cochran-Mantel-Haenszel; Stratified difference = -1.6, 95% CI 2-sided [-8.3 to 5.9] — The weighted average of the treatment differences across the strata with CMH weights
Statistical Analysis 2: Comparison: Placebo vs GED-0301 160 mg / GED-0301 40 mg; Test type: Superiority; p = 0.2221, Cochran-Mantel-Haenszel; Stratified difference = -2.0, 95% CI 2-sided [-8.7 to 5.1] — The weighted average of the treatment differences across the strata with the CMH weights
Statistical Analysis 3: Comparison: Placebo vs GED-0301 160 mg / GED-0301 160 mg 4 Week Alt; Test type: Superiority; p = 0.2578, Cochran-Mantel-Haenszel; Stratified difference = -2.0, 95% CI 2-sided [-8.7 to 5.6] — The weighted average of the treatment differences across the strata with the CMH weights

10. Secondary Outcome: The Number of Participants Who Experienced Treatment Emergent Adverse Events (TEAE) From Week 0 to Week 52
Description: A TEAE was defined as any adverse event (AE) occurring or worsening on or after the first treatment of GED-0301 and up to 28 days after the last GED-0301 dose or the last follow-up date, whichever occurred earlier. A serious AE = any AE which results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; constitutes an important medical event.
Time Frame: From the first day of GED-0301 until 28 days after the last dose of investigational product (IP); maximum treatment duration was 52.6 weeks
Population: The safety population consisted of all participants who were randomized and received at least 1 dose of IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GED-0301 160 mg / GED-0301 40 mg 4 Week Alt | GED-0301 160 mg / GED-0301 40 mg | GED-0301 160 mg / GED-0301 160 mg 4 Week Alt
Number analyzed (Participants) | 174 | 176 | 176 | 175
Participants
  Any TEAE | 124 | 128 | 129 | 113
  Any IP-Related TEAE | 31 | 35 | 30 | 20
  Any Severe TEAE | 14 | 22 | 21 | 15
  Any Serious TEAE (SAE) | 16 | 28 | 22 | 15
  Any Serious IP-Related TEAE | 3 | 2 | 2 | 0
  Any TEAE Leading to IP Withdrawal | 11 | 15 | 16 | 12
  Any TEAE Leading to IP Interruption | 4 | 4 | 5 | 4
  Any TEAE Leading to Death | 0 | 0 | 1 | 1

11. Secondary Outcome: The Number of Participants Who Discontinued IP Due to an Treatment Emergent Adverse Events
Description: A TEAE was defined as any AE occurring or worsening on or after the first dose of GED-0301 and up to 28 days after the last GED-0301 dose or the last follow-up date, whichever occurred earlier. A serious AE = any AE which results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; constitutes an important medical event. The severity of AEs was assessed by the investigator and based on the following scale: Mild = asymptomatic or mild symptoms; clinical or diagnostic observations only; Moderate = Symptoms cause moderate discomfort; Severe (could be non-serious or serious) = symptoms causing severe discomfort/pain.
Time Frame: From the first day of GED-0301 until 28 days after the last dose of IP; maximum treatment duration was 52.6 weeks
Population: The safety population consisted of all participants who were randomized and received at least 1 dose of IP
Measure: Number; unit: participants
Arm/Group | Placebo | GED-0301 160 mg / GED-0301 40 mg 4 Week Alt | GED-0301 160 mg / GED-0301 40 mg | GED-0301 160 mg / GED-0301 160 mg 4 Week Alt
Number analyzed (Participants) | 174 | 176 | 176 | 175
participants | 11 | 15 | 16 | 12

12. Primary Outcome: The Percentage of Participants Who Achieved a Clinical Remission at Week 12
Description: Clinical remission is defined as a Crohn's Disease Activity Index (CDAI) score < 150. The Crohn's Disease Activity Index is used to quantify the signs and symptoms of Crohn's disease and the affect on patient's quality of life. It consists of 8 variables which include patient reported outcomes over a 7 day period and physician assessments which are scored numerically and weighted. Scores range from 0 to 600, with the most severe disease defined >450.
Time Frame: Week 12
Population: ITT population; includes participants who had either completed that timepoint visit or discontinued at any time due to reasons other than study terminated by sponsor; the Non-responder Imputation (NRI)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | GED-0301 160 mg / GED-0301 40 mg 4 Week Alt | GED-0301 160 mg / GED-0301 40 mg | GED-0301 160 mg / GED-0301 160 mg 4 Week Alt
Number analyzed (Participants) | 160 | 162 | 164 | 157
Percentage of Participants | 25.0 [18.9 to 32.2] | 25.3 [19.2 to 32.5] | 21.3 [15.8 to 28.2] | 21.7 [15.9 to 28.7]
Statistical Analysis 1: Comparison: Placebo vs GED-0301 160 mg / GED-0301 40 mg 4 Week Alt; Test type: Superiority; p = 0.9141, Cochran-Mantel-Haenszel; Stratified Difference = 0.5, 95% CI 2-sided [-8.9 to 10.0] — The weighted average of the treatment differences across the strata with the Cochran-Mantel-Haenszel (CMH) weights
Statistical Analysis 2: Comparison: Placebo vs GED-0301 160 mg / GED-0301 40 mg; Test type: Superiority; p = 0.4286, Cochran-Mantel-Haenszel; Stratified Difference = -3.6, 95% CI 2-sided [-12.8 to 5.6] — The weighted average of the treatment differences across the strata with the CMH weights
Statistical Analysis 3: Comparison: Placebo vs GED-0301 160 mg / GED-0301 160 mg 4 Week Alt; Test type: Superiority; p = 0.5591, Cochran-Mantel-Haenszel; Stratified Difference = -2.7, 95% CI 2-sided [-12.0 to 6.6] — The weighted average of the treatment differences across the strata with the CMH weights

ADVERSE EVENTS:
Time Frame: From day 1 of GED-0301 until 28 days after the last dose of IP as well as those SAEs made known to the Investigator at any time thereafter that are suspected of being related to IP.
Description: Maximum treatment duration was 52.6 weeks
Arm/Group | Placebo | GED-0301 160 mg / GED-0301 40 mg 4 Week Alt | GED-0301 160 mg / GED-0301 40 mg | GED-0301 160 mg / GED-0301 160 mg 4 Week Alt
All-Cause Mortality (participants affected / at risk) | 0/174 | 0/176 | 1/176 | 1/175
Serious Adverse Events (participants affected / at risk) | 16/174 | 28/176 | 22/176 | 15/175
Other Adverse Events (participants affected / at risk) | 78/174 | 72/176 | 74/176 | 63/175
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=174) | GED-0301 160 mg / GED-0301 40 mg 4 Week Alt (N=176) | GED-0301 160 mg / GED-0301 40 mg (N=176) | GED-0301 160 mg / GED-0301 160 mg 4 Week Alt (N=175)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
ABDOMINAL ADHESIONS (Gastrointestinal disorders) | 0 | 1 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 | 1 | 1 | 2
ANAL FISSURE (Gastrointestinal disorders) | 0 | 1 | 0 | 0
ANAL FISTULA (Gastrointestinal disorders) | 0 | 2 | 2 | 0
COLITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 1
CROHN'S DISEASE (Gastrointestinal disorders) | 4 | 9 | 8 | 5
ENTEROVESICAL FISTULA (Gastrointestinal disorders) | 0 | 0 | 0 | 1
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 | 0 | 1 | 0
ILEAL STENOSIS (Gastrointestinal disorders) | 0 | 1 | 0 | 0
INTESTINAL STENOSIS (Gastrointestinal disorders) | 0 | 1 | 0 | 0
LARGE INTESTINAL STENOSIS (Gastrointestinal disorders) | 1 | 0 | 0 | 0
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 0 | 1 | 0 | 0
MELAENA (Gastrointestinal disorders) | 1 | 0 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 0 | 1 | 0 | 0
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 | 0 | 0 | 1
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 2 | 1 | 2
VOMITING (Gastrointestinal disorders) | 2 | 0 | 0 | 1
ASTHENIA (General disorders) | 0 | 1 | 0 | 0
DRUG WITHDRAWAL SYNDROME (General disorders) | 0 | 0 | 0 | 1
FATIGUE (General disorders) | 0 | 1 | 0 | 0
PYREXIA (General disorders) | 0 | 0 | 1 | 0
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 | 1 | 0 | 0
HEPATIC VEIN THROMBOSIS (Hepatobiliary disorders) | 0 | 0 | 1 | 0
HEPATITIS (Hepatobiliary disorders) | 0 | 1 | 0 | 0
ABDOMINAL ABSCESS (Infections and infestations) | 0 | 0 | 1 | 0
ANAL ABSCESS (Infections and infestations) | 1 | 1 | 1 | 0
CELLULITIS (Infections and infestations) | 1 | 0 | 0 | 1
EPSTEIN-BARR VIRUS INFECTION (Infections and infestations) | 1 | 0 | 0 | 0
GASTROENTERITIS (Infections and infestations) | 0 | 1 | 0 | 0
GASTROENTERITIS NOROVIRUS (Infections and infestations) | 0 | 1 | 0 | 0
HERPES SIMPLEX OESOPHAGITIS (Infections and infestations) | 0 | 1 | 0 | 0
HERPES ZOSTER (Infections and infestations) | 0 | 0 | 1 | 0
PNEUMONIA (Infections and infestations) | 0 | 0 | 1 | 0
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 0 | 0 | 1 | 0
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
PROCEDURAL INTESTINAL PERFORATION (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
WEIGHT DECREASED (Investigations) | 0 | 0 | 0 | 1
MALNUTRITION (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
CERVIX NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
NEUROENDOCRINE TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
HEADACHE (Nervous system disorders) | 0 | 1 | 0 | 0
SCIATICA (Nervous system disorders) | 1 | 0 | 0 | 0
DEVICE DISLOCATION (Product Issues) | 1 | 0 | 0 | 0
ALCOHOLISM (Psychiatric disorders) | 0 | 0 | 1 | 0
STRESS URINARY INCONTINENCE (Renal and urinary disorders) | 1 | 0 | 0 | 0
PERINEAL DISORDER (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
ACUTE FEBRILE NEUTROPHILIC DERMATOSIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
PSORIASIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
PYODERMA GANGRENOSUM (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=174) | GED-0301 160 mg / GED-0301 40 mg 4 Week Alt (N=176) | GED-0301 160 mg / GED-0301 40 mg (N=176) | GED-0301 160 mg / GED-0301 160 mg 4 Week Alt (N=175)
ABDOMINAL PAIN (Gastrointestinal disorders) | 19 | 20 | 14 | 15
CROHN'S DISEASE (Gastrointestinal disorders) | 15 | 14 | 14 | 15
DIARRHOEA (Gastrointestinal disorders) | 0 | 10 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 12 | 9 | 10 | 9
PYREXIA (General disorders) | 10 | 13 | 14 | 0
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 15 | 18 | 14 | 16
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 15 | 20 | 23 | 25
BACK PAIN (Musculoskeletal and connective tissue disorders) | 9 | 0 | 0 | 0
HEADACHE (Nervous system disorders) | 15 | 10 | 12 | 9

LIMITATIONS AND CAVEATS:
Following a recommendation by the DMC, this study was terminated early by the sponsor on 19 Oct 2017 due to a lack of emerging benefit; no emergent safety findings were noted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is > 1 year since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to 90 additional days. Investigator must delete confidential information before submission and defer publication to permit patent applications.

DOCUMENTS (2):
  • Study Protocol (2017-08-15): https://cdn.clinicaltrials.gov/large-docs/93/NCT02596893/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/93/NCT02596893/SAP_001.pdf